CLINICAL TRIAL: NCT00213616
Title: Bilateral Laryngeal Paralysis Reinnervation. Speech and Ventilatory Results Analysis
Brief Title: Bilateral Laryngeal Paralysis Reinnervation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1999/141/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Vocal Cord Paralysis
Keywords: bilateral vocal cord paralysis; reinnervation; phrenic nerve
MeSH Terms: conditions — Vocal Cord Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: surgical reinnervation — laryngeal reinnervation with a phrenic nerve root

SUMMARY:
Bilateral laryngeal reinnervation induces a rise in laryngeal resistance and speech alteration. The aim of this study is to propose laryngeal reinnervation by a phrenic nerve root to patients with bilateral laryngeal paralysis.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral laryngeal paralysis without any amelioration for six months

Exclusion Criteria:

* Laryngeal paralysis more than 3 years
* Arycricoideus ankylostosis
* Pacemaker
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
LARYNGEAL REINNERVATION | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean Paul Marie, MD, PHD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France